CLINICAL TRIAL: NCT00442871
Title: An Open-Label, Non-Randomized Pharmacokinetic and Safety Study of a Single Oral Dose of 50 mg Eltrombopag in Healthy Subjects and in Subjects With Mild, Moderate, or Severe Renal Impairment
Brief Title: Study Of SB-497115 in Healthy Subjects and Subjects With Mild, Moderate or Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRA104412
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: Renal Impairment,; chronic immune thrombocytopenia purpura,; thrombocytopenia,; chemotherapy induced thrombocytopenia
MeSH Terms: conditions — Purpura; Renal Insufficiency; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag 50 mg oral (single dose)
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — eltrombopag 50 mg oral

SUMMARY:
The main purpose of this study is to compare how one 50 mg tablet of SB-497115 is broken down in the body by healthy subjects versus subjects with mild, moderate or severe kidney problems. The study is also being done to 1) check on how well the study drug is tolerated by healthy subjects versus those with liver problems and 2) to check if liver impairment affects how the study drug binds to protein in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or have renal impairment
* Females (the following requirement applies only if able to have children): agree to doctor approved birth control methods, or partner has had a vasectomy
* Negative drug, alcohol, and HIV tests.

Exclusion Criteria:

* Taking a medication or therapy not approved by the study doctor
* Rapidly changing kidney function
* Drug or alcohol abuse within past 6 months
* Used an investigational drug in the past 30 days
* Females who are pregnant or nursing
* Have active hepatitis B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-09-28 (Actual); Primary Completion 2008-01-03 (Actual); Study Completion 2008-01-03 (Actual)

PRIMARY OUTCOMES:
Plasma levels and protein binding of eltrombopag | at Day 1 to Day 6.
  plasma levels/protein binding for eltrombopag

SECONDARY OUTCOMES:
Safety will be assessed by: -eye exam | at Screening, Day -1, & followup
  eye exam safety findings
adverse assessment | Day 1 to followup
  Adverse event review
clinical labs, vital signs, & 12-lead electrocardiograms done | all days but Day 4
  Clinical labs, vital signs and 12 lead electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Saint Paul, Minnesota

REFERENCES:
- [Background] Bauman JW, Vincent CT, Peng B, Wire MB, Williams DD, Park JW. Effect of hepatic or renal impairment on eltrombopag pharmacokinetics. J Clin Pharmacol. 2011 May;51(5):739-50. doi: 10.1177/0091270010372106. Epub 2010 Jul 27. PMID 20663991
- See also: Results for study TRA104412 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/TRA104412?search=study&search_terms=TRA104412#rs